CLINICAL TRIAL: NCT00951743
Title: Safety and Efficacy of ADAPTAVIR's Ability to Eliminate Treatment-Resistant Infectious Virus in the Blood Cellular Reservoir (PBMCs) of HIV Patients With Suppressed Plasma Viral Load.
Brief Title: Safety and Efficacy of ADAPTAVIR's Ability to Eliminate Treatment-Resistant Infectious Virus in Peripheral Blood Mononuclear Cells (PBMCs)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rapid Laboratories Inc. (Other)
Responsible Party: Richard Elion/Prinicpal Investigator, Whitman Walker Clinic
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAPID Laboratories 001
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
Keywords: AIDS; HIV; mDAPTA
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — D-Ala-peptide T-amide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Adaptavir Treatment (Experimental): MDAPTA (Adaptavir) will be administered intranasally at 0.01 mg twice per day. Individuals with plasma viral load (PCR Roche Amplicor Ultrasensitive assay) less than 200 copies/mL, sustained for the previous 90 days, with CD4>350 cells/mm3 will be eligible to participate.
  Interventions: Drug: Adaptavir (monomeric DAPTA)
- Placebo (Placebo Comparator): Placebo will be administered intranasally at 0.01 mg twice per day. Individuals with plasma viral load (PCR Roche Amplicor Ultrasensitive assay) less than 200 copies/mL, sustained for the previous 90 days, with CD4>350 cells/mm3 will be eligible to participate.
  Interventions: Drug: Adaptavir (monomeric DAPTA)

INTERVENTIONS:
Drug: Adaptavir (monomeric DAPTA) — Intranasal (IN) Solution: 20 mL of solution in a 20 mL polyethylene screw top vial to which a metered sprayer is adapted. Each spray releases approximately 0.1 0.12 mL.
  Available strength - 0.01mg/mI (active study medication), or no mDAPTA (placebo study medication), in water containing 0.25% benzyl alcohol as preservative and 250 mM mannitol (GRAS) to achieve isotonicity.
  Individuals in this study will be randomized to receive mDAPTA or placebo and be instructed to administer four metered nasal spray applications two times a day, in the morning, and in the evening, as close to 12 hours after the morning dose as practical. The planned daily dose of mDAPTA is 8 μg/day.
  Other Names: Adaptavir; Monomeric DAPTA; DAPTA -D ala Peptide T

SUMMARY:
This is a 24 week placebo controlled, double-blind, 2-arm study of ADAPTAVIR, Monomeric Dala1-peptide T-amide (mDAPTA) compared to placebo, in HIV infected individuals with suppressed plasma viral loads < 200 copies/ml by highly active antiretroviral therapy (HAART) treatment for at least 3 months prior to entry with at least 6 continuous months of HAART treatment preceding entry. 20 treatment and 20 placebo individuals will be enrolled in each arm. The study duration is 24 weeks on placebo or mDAPTA administered intranasally at 0.01 mg two times a day.

The main (intent to treat) analysis is planned for the 24 week endpoint. The virological outcomes of interest in the present study are infectious virus recoverable from cellular (PBMC) sources and cellular viral mRNA and DNA copy numbers. Immune outcomes (plasma cytokines) associated with HIV disease, HIV replication, or immune function will be studied.

DETAILED DESCRIPTION:
A primary objective of this study is to assess the safety and toxicity of mDAPTA (Adaptavir) in HIV infected individuals with suppressed viral loads with HAART treatment and assess the proportion of study participants achieving PMBC viral culture negative status at 24weeks. PMBC viral culture status is a direct measurement of treatment resistant, residual, active HIV replication in the peripheral blood mononuclear cells. We hypothesize this proportion will be significantly greater in the treatment arm relative to the placebo arm (the odds of achieving this endpoint are significantly greater in mDAPTA- than in placebo-treated participants).

Secondary Endpoints (all analyzed as odds ratios) are to determine

* The proportion of study participants achieving (0.5 log10) decrease in quantitative viral mRNA in PBMCs will be significantly greater in the treatment arm relative to the placebo arm.
* The proportion of study participants achieving (0.5 log10) decrease in quantitative viral DNA in PBMCs will be significantly greater in the treatment arm relative to the placebo arm.
* The proportion of study participants whose plasma viral loads were greater than 200 copies/ml on two successive measurements 6 weeks apart will be significantly greater in the placebo arm relative to the treatment arm.

Immunological outcome hypotheses, based on 24-week data

* The proportion of study participants achieving at least greater than 50% decrease in the inflammatory cytokines TNFa, IL-10, IL-8 or IL-6 will be significantly greater in the treatment arm relative to the placebo arm.
* The proportion of study participants achieving at least greater than 50% increase in the cytokines IL-2, IL-10, IL-12, IL-13 and IFNa will be significantly greater in the treatment arm relative to the placebo arm.
* The proportion of study participants achieving at least an increase in CD4 T cells will be significantly greater in the treatment arm relative to the placebo arm.
* The proportion of study participants whose viral load becomes greater than 200 copies/ml will be significantly greater in the placebo arm relative to the treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. HIV positive, male or female of any race and at least 18 years of age.
2. Must have received continuous currently acceptable anti-retroviral therapy ("HAART"; highly active antiviral therapy) for at least six months prior to entry.
3. Must have HIV-1 plasma viral load RNA (PCR or bDNA) < 200 copies/mL for 90 days prior to randomization in this study.
4. Women of childbearing potential must have a negative pregnancy test at screening prior to randomization in this study. Upon randomization, these women must agree to use methods of birth control or abstinence to prevent pregnancy.
5. Must have a sustained CD4+ cell count > 350 cells/mm3 for 90 days prior to randomization in this study.
6. Must be considered clinically stable, in the opinion of the investigator, at the time of entry into the study.

Exclusion Criteria:

1. Expected to require adjustment to their antiretroviral therapy during screening or within 8 weeks after initiating mDAPTA therapy.
2. Current participation in other clinical trials with investigational drugs.
3. Use of any investigational agents including immunomodulatory agents (GM CSF, interferon, interleukin etc.) within 60 days prior to study entry.
4. Use of any vaccine, including for Influenza (killed or live), Pneumovax etc., within 60 days of initiating therapy with mDAPTA.
5. Use or anticipated use of immunosuppressive therapy, including chemotherapy during participation in the study.
6. Alcohol or substance abuse which, in the opinion of the investigator, would interfere with patient compliance or safety.
7. Study participants with an active opportunistic infection or malignancy.
8. Pregnant or breastfeeding.
9. Any condition or history of any illness which, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drugs to the participant.
10. Participants who previously received treatment with DAPTA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-05 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
To assess the safety & toxicity of mDAPTA in HIV infected individuals with suppressed viral loads on HAART treatment & assess the proportion of study participants achieving PMBC viral culture negative status at 24weeks. | 6 months with 2 month follow up

SECONDARY OUTCOMES:
Virological and Immunological outcome measures | 6 months with 2 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Richard Elion, MD, Principal Investigator — Whitman Walker clinic
Locations (1):
- Whitman Walker Clinic, Washington D.C., District of Columbia, United States